CLINICAL TRIAL: NCT03462849
Title: Expiratory Fow Assessment in ARDS Patients
Brief Title: Expiratory Flow Limitation Assessment
Acronym: FLAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0595; 2017-A02557-46 (Other: ANSM)
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; expiratory flow limitation; trans-pulmonary pressure; airway closure
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with EFL at PEP 5 (Other): Patients with EFL at PEP 5 at the time of inclusion either in supine or semi-recumbent position
  Interventions: Other: increase in positive end expiratory pressure
- Patients with no EFL at PEP 5 (Other): Patients with no EFL at PEP 5 at the time of inclusion in both supine and semi-recumbent positions
  Interventions: Other: increase in positive end expiratory pressure

INTERVENTIONS:
Other: increase in positive end expiratory pressure — increase in positive end expiratory pressure from 5 to 10 then 15 cmH2O then at the value for trans pulmonary end expiratory pressure amounting to 3 cmH2O

SUMMARY:
This study intended to assess the expiratory flow limitation (EFL) during tidal breath in patients intubated in intensive care unit (ICU) for moderate or severe acute respiratory distress syndrome (ARDS). EFL is defined as the lack of increase in expiratory flow in response to an increase in alveolar-to-atmospheric pressure gradient. It reflects airway closure. Early studies have been done using the Negative expiratory pressure (NEP) technique, which is no longer available. We proposed in present study a new method, which consists of diverting manually the expiratory flow to the atmosphere by-passing the expiratory valve. We aimed at assessing EFL at positive expiratory pressure (PEP) 5 cmH2O in semi-recumbent then in supine position together with measurement of trans-pulmonary pressure and regional lung ventilation. Higher PEP levels will be tested, namely 10, 15 and a trans-pulmonary PEP of 3 cmH2O, in semi-recumbent position.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or more in age
* moderate to severe ARDS according to the Berlin definition : Intubated (or tracheotomized) and mechanically ventilated in the ICU
* no pregnancy
* informed consent from the next of kin

Exclusion Criteria:

* Contra-indication to PEP > 5 cmH2O
* extracorporeal membrane oxygenation (ECMO)
* chest tube
* mean arterial pressure < 65 mmHg
* Contra-indication to oesophageal device
* underlying disease fatal in less than one year
* active therapy limitation
* under guardian
* refusal to participate
* not affiliated to insurance regimen
* speaking barrier of the next of kin
* investigator not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
EFL at PEP 5 cmH2O | at inclusion
  A Fleish 2 pneumotachograph and a port to measure airway pressure are attached at the Y piece of the ventilator circuit and connected to a Biopac 150. At the end of inspiration the air is expelled to the atmosphere upstream the expiratory valve. The flow volume loop at baseline and that during the manoeuver are plotted and patients classified as EFL or not EFL (NFL). Measurements are taken in semi-recumbent then after 5 minutes in supine position.

SECONDARY OUTCOMES:
Trans-pulmonary pressure at end expiratory at PEP 5 | at inclusion
  After insertion of esophageal balloon together with pneumotachograph and port for airway pressure trans-pulmonary pressure (airway-esophageal pressure) is measured after a 3-sec end-expiratory pause in semi-recumbent and then after 5 minutes in supine position
Trans-pulmonary pressure at end expiratory at PEP 10 in EFL and NFL patients | 15 minutes after PEP set to 10 cm H2O
  PEP is increased to 10 cmH2O and 15 minutes later trans-pulmonary pressure is measured after a 3-sec end-expiratory pause in semi-recumbent position
Lung compliance at PEP 10 in EFL and NFL patients | 15 minutes after PEP set to 10 cm H2O
  PEP is increased to 10 cmH2O and 15 minutes later lung compliance is measured after a 3-sec end-expiratory pause in semi-recumbent position
lung ventilation distribution at PEP 10 in EFL and NFL patients | 15 minutes after PEP set to 10 cm H2O
  PEP is increased to 10 cmH2O and 15 minutes later lung ventilation is measured by using electrical impedance tomography (EIT) in semi-recumbent position (an EIT belt having been inserted together with the previous measurement devices).
Transcutaneous oxygen saturation (SpO2) at PEP 10 in EFL and NFL patients | 15 minutes after PEP set to 10 cm H2O
  PEP is increased to 15cmH2O and 15 minutes later SpO2 is read from the vital functions monitoring device and SpO2/FIO2 computed
Trans-pulmonary pressure at end expiratory at PEP 15 in EFL and NFL patients | 15 minutes after PEP set to 15 cm H2O
  PEP is increased to 15 cmH2O and 15 minutes later trans-pulmonary pressure is measured after a 3-sec end-expiratory pause in semi-recumbent position
Lung compliance at PEP 15 in EFL and NFL patients | 15 minutes after PEP set to 15 cm H2O
  PEP is increased to 15 cmH2O and 15 minutes later lung compliance is measured after a 3-sec end-expiratory pause in semi-recumbent position
lung ventilation distribution at PEP 15 in EFL and NFL patients | 15 minutes after PEP set to 15 cm H2O
  PEP is increased to 15 cmH2O and 15 minutes later lung ventilation is measured by using electrical impedance tomography (EIT) in semi-recumbent position (an EIT belt having been inserted together with the previous measurement devices).
transcutaneous oxygen saturation (SpO2) at PEP 15 in EFL and NFL patients | 15 minutes after PEP set to 15 cm H2O
  PEP is increased to 15 cmH2O and 15 minutes later SpO2 is read from the vital functions monitoring device and SpO2/FIO2 computed.
Trans-pulmonary pressure at end expiratory at PEP to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O in EFL and NFL patients | 15 minutes after PEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O
  PEP is set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O and 15 minutes later trans-pulmonary pressure is measured after a 3-sec end-expiratory pause in semi-recumbent position
Lung compliance at PEP to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O in EFL and NFL patients | 15 minutes after PEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O
  PEP is set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O and 15 minutes later lung compliance is measured after a 3-sec end-expiratory pause in semi-recumbent position
lung ventilation distribution at PEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O in EFL and NFL patients | 15 minutes after PEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O
  PEP is set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O and 15 minutes later lung ventilation is measured by using electrical impedance tomography (EIT) in semi-recumbent position (an EIT belt having been inserted together with the previous measurement devices).
Transcutaneous oxygen saturation (SpO2) at PEEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O in EFL and NFL patients | 15 minutes after PEEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O
  PEEP is increased to 15 cmH2O and 15 minutes later SpO2 is read from the vital functions monitoring device and SpO2/FIO2 computed.
lung recruitment at PEEP 10 in EFL and NFL patients | 15 minutes after PEEP set to 10 cm H2O
  PEEP is increased to 10 cmH2O and 15 minutes later lung recruitment is measured between PEEP 10 and PEEP 5 (in each body position) from volume-pressure curves recorded at PEEP 10 and PEEP 5. The lung recruitment is the change in lung volume for a given pressure (higher PEEP and 20 cmH2O)
lung recruitment at PEEP 15 in EFL and NFL patients | 15 minutes after PEEP set to 15 cm H2O
  PEEP is increased to 15 cmH2O and 15 minutes later lung recruitment is measured between PEEP 15 and PEEP 5 (in each body position) from volume-pressure curves recorded at PEEP 15 and PEEP 5. The lung recruitment is the change in lung volume for a given pressure (higher PEEP and 20 cmH2O)
lung recruitment at PEEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O in EFL and NFL patients in EFL and NFL patients | 15 minutes after PEEP set to 15 cm H2O
  PEEP is increased to PEEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O and 15 minutes later lung recruitment is measured between PEEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O and PEEP 5 (in each body position) from volume-pressure curves recorded at PEEP set to reach Trans-pulmonary pressure at end expiratory =+3 cmH2O and PEEP 5. The lung recruitment is the change in lung volume for a given pressure (higher PEEP and 20 cmH2O)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Guerin, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble
  - Hôpital de la Croix Rousse, Lyon

REFERENCES:
- [Result] Guerin C, Terzi N, Galerneau LM, Mezidi M, Yonis H, Baboi L, Kreitmann L, Turbil E, Cour M, Argaud L, Louis B. Lung and chest wall mechanics in patients with acute respiratory distress syndrome, expiratory flow limitation, and airway closure. J Appl Physiol (1985). 2020 Jun 1;128(6):1594-1603. doi: 10.1152/japplphysiol.00059.2020. Epub 2020 Apr 30. PMID 32352339